CLINICAL TRIAL: NCT04687878
Title: Evaluating the Effect of Intranasal Insulin Administration on Motor and Non-motor Symptoms in Parkinson's Disease Patients; a Randomized Double-blinded Placebo-controlled Clinical Trial
Brief Title: The Effect of Intranasal Insulin on Motor and Non-motor Symptoms in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: dr.dargahi (Other)
Responsible Party: Sponsor-Investigator, dr.dargahi, Associate professor, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SBMU.PHNS.REC.1398.094
Record Dates: First submitted 2020-12-28; First posted 2020-12-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Insulin; Intranasal; Motor symptoms; Non-motor symptoms
MeSH Terms: conditions — Parkinson Disease; Insulin Resistance | interventions — Insulin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin (Experimental): Regular Insulin, 20 IU twice a day, intranasally, every day for 12 weeks
  Interventions: Drug: Insulin
- Placebo (Placebo Comparator): Normal saline, twice a day, intranasally, every day for 12 weeks
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Insulin — 20 IU twice a day, intranasally, every day for 12 weeks
  Other Names: Insulin regular
  Arms: Insulin
Drug: Normal saline — twice a day, intranasally, every day for 12 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of intranasal insulin on motor and non-motor symptoms of patients with Parkinson's disease over a 12-week period.

DETAILED DESCRIPTION:
This study is a single-center, parallel and double-blind study. Patients with Parkinson's disease referred to Movement Clinic of Shohada-e-Tajrish Hospital will randomly receive intranasal placebo or insulin, every day, twice a day for 12 weeks. Motor and non-motor symptoms will be evaluated in four time points; baseline, 4, 8 and 12 weeks after treatments. Primary outcome is motor symptoms (MDS-UPDRS; part III, IV), and secondary outcomes are motor (gait balance) and non-motor (MDS-UPDRS part I, II, cognition, depression, anxiety and fatigue) symptoms. Patients, researchers (physicians, outcome assessors) and data analysts are blinded.

ELIGIBILITY:
Inclusion Criteria:

* Man and woman over 17 years old
* Patient with Parkinson's disease according to UK Parkinson's Disease Society Brain Bank Diagnostic Criteria
* Provide written informed consent to participate in the study.
* Understand that they may withdraw their consent at any time.

Exclusion Criteria:

* Pregnant and lactating women
* Patients with diabetes and taking anti-hyperglycemic drugs
* Patients with other neurodegenerative diseases like multiple system atrophy, Huntington's, Wilson's disease, Alzheimer's, Amyotrophic lateral sclerosis (ALS), progressive supranuclear palsy, etc.
* Patients who cannot walk for more than one minute without help
* A history of allergic reaction to insulin
* The presence of inflammation of nasal cavity that may prevents absorption of insulin

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III, IV | Base line, 4, 8 and 12 weeks after intervention
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III, IV assess the motor signs of Parkinson's Disease; higher score means more severity of the motor symptoms.

SECONDARY OUTCOMES:
Changes in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I, II | Base line, 4, 8 and 12 weeks after intervention
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I, II assess the non motor signs of PD; higher score means more severity of the symptoms.
Disease severity | Base line, 4, 8 and 12 weeks after intervention
  The modified Hoehn and Yahr Scale (HY) is used to assess severity of Parkinson's Disease. The scale ranges from 1 to 5. The lower score indicates better outcome.
Risk of Falling | Base line, 4, 8 and 12 weeks after intervention
  Tinetti Balance Assessment Tool indicates the risk of falling, higher scores is indicative of low risk for falling.
Cognitive score | Base line, 4, 8 and 12 weeks after intervention
  The Montreal Cognitive Assessment (MoCA) scores range between 0 and 30 with higher scores indicative of better cognitive performance.
Depression score | Base line, 4, 8 and 12 weeks after intervention
  Beck's Depression Inventory II (BDI-II) scores range between 0 and 63; higher scores is indicative of more severe depression.
Anxiety score | Base line, 4, 8 and 12 weeks after intervention
  Beck Anxiety Inventory (BAI) scores range between 0 and 63; higher scores is indicative of more anxiety.
Fatigue score | Base line, 4, 8 and 12 weeks after intervention
  Fatigue Severity Scale (FSS) scores range between 0 and 7; higher scores is indicative of severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Dargahi, PharmD/PhD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mehri Salari, MDFellowship, Principal Investigator — Shahid Beheshti University of Medical Sciences; Abolhassan Ahmadiani, PharmD/PhD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Neda Valian, PhD, Study Director — Shahid Beheshti University of Medical Sciences; Leila Mohaghegh Shalmani, PharmD/PhD, Study Chair — Shahid Beheshti University of Medical Sciences; Helia Ashourizadeh, Intern, Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University of Medical Sciences, Shohada-e-Tajrish Hospital, Tehran, Iran